CLINICAL TRIAL: NCT03564782
Title: Examining Oncolytic Poliovirus Bioactivity in Tumor Tissue After Intratumoral Administration of PVSRIPO in Women With Invasive Breast Cancer
Brief Title: Examining Bioactivity of PVSRIPO in Invasive Breast Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Istari Oncology, Inc. (Industry)
Collaborators: Duke University (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00085352; W81XWH-16-1-0354 (Other Grant/Funding Number: US Department of Defense (DoD))
Record Dates: First submitted 2018-06-10; First posted 2018-06-21 (Actual); Results first posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2023-06

CONDITIONS: Invasive Breast Cancer
Keywords: PVSRIPO; Invasive Breast Cancer

STUDY DESIGN:
Intervention Model Description: All subjects will receive intratumoral injection of the study drug PVSRIPO at a dose of 1x10^8 TCID50 (tissue culture infectious dose). On Day 14 after injection, subjects will undergo standard-of-care surgical resection of PVSRIPO-treated tumor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PVSRIPO (Experimental): Polio vaccine booster will be administered 1 week prior to PVSRIPO injection. On the day of PVSRIPO injection (Day 0), a pre-treatment biopsy is obtained. PVSRIPO in injected into the tumor mass at a dose of 1x10^8 TCID50. On day 14, women will undergo standard-of-care surgical resection of PVSRIPO-treated tumor.
  Interventions: Biological: PVSRIPO

INTERVENTIONS:
Biological: PVSRIPO — The live, attenuated, oral (Sabin), serotype 1 poliovirus vaccine booster will be administered 1 week before PVSRIPO injection. The study drug, PVSRIPO, is the live attenuated, oral (Sabin) serotype 1 poliovirus vaccine containing a heterologous internal ribosomal entry site (IRES) derived from the human rhinovirus type 2 (HRV2). It will be given at a dose of 1x10^8 TCID50 (tissue culture infectious dose) directly into the breast tumor.

SUMMARY:
This is a pilot study to examine PVSRIPO bioactivity in tumor tissue after intratumoral administration of PVSRIPO in women with invasive breast cancer.

DETAILED DESCRIPTION:
The study drug PVSRIPO is the live attenuated, oral (Sabin) serotype 1 poliovirus vaccine containing a heterologous internal ribosomal entry site (IRES) derived from the human rhinovirus type 2 (HRV2). The purpose of this pilot study is to examine PVSRIPO bioactivity in tumor tissue after intratumoral administration of PVSRIPO in women with invasive breast cancer. The hypothesis is that administration of PVSRIPO in the tumor causes inflammation, which stimulates innate and adaptive immune activation in invasive breast cancer. Enrollment target will include six women with invasive breast cancer. Women with stage II-IV invasive breast cancer with at least 1 cm of residual tumor after chemotherapy and scheduled for standard of care surgery will be eligible.

The objective of the study is to investigate PVSRIPO-mediated inflammation and immunity in women invasive breast cancer. The primary exploratory objective is to describe the change in the amount of tumor infiltrating immune cells in tumor tissue pre- and post-injection of PVSRIPO by H&E (Haemotoxylin and Eosin).

Other exploratory objectives are: 1.) to examine tumor tissue pre- and post-injection of PVSRIPO for inflammatory and immune signature using arrays, CD155 expression by immunohistochemistry (IHC), immune cell infiltrate by IHC and tumor infiltrating immune cells using flow cytometry (post-injection only); and 2) To examine blood for inflammatory and immune signature using arrays, immune cell composition (antigen presenting cells, B cells and T cells), T cell activation by flow cytometry and B cell activation by ELISA and peptide arrays. Blood will be collected on day -7 (before polio vaccine booster), day 0 (before PVSRIPO injection), day 2 (after PVSRIPO), day 14 (after PVSRIPO before surgery), and in follow-up at months 1 and 6 post-PVSRIPO.

ELIGIBILITY:
This pilot study will include women with stage II-IV ER/PR/HER2 negative (triple negative) breast cancer scheduled to undergo surgical resection.

Inclusion Criteria:

* Age ≥ 18 years
* Confirmation of invasive breast cancer including any of the following:

  * Triple-negative breast cancer defined as receptor status being estrogen receptor expression ≤ 10%, progesterone receptor expression ≤ 10%, and HER2/Neu expression by IHC 0 or 1+, or 2+ with fluorescence in situ hybridization confirming no amplification of HER2 on a pretreatment tumor sample.
  * Hormone positive breast cancer defined as receptor status being estrogen receptor expression > 10%, progesterone receptor expression > 10% prior to initiation of chemotherapy.
  * HER2+ breast cancer defined as HER2/Neu expression by IHC 3+ or fluorescence in situ hybridization confirming amplification of HER2 on a pretreatment tumor sample prior to initiation of chemotherapy. HER2+ and hormone positive (ie triple positive) breast cancers are included in this study.
* Stage II-III invasive breast cancer with ≥ 1 cm of residual tumor based on MRI, mammogram, ultrasound, or breast clinical exam as SOC after completion of neoadjuvant chemotherapy, OR Stage IV BC with ≥ 1 cm locally recurrent disease (i.e. chest wall recurrence only)
* ECOG ≤ 1
* Hemoglobin ≥ 9.0 g/dl, ANC ≥ 1,500 cells/µl, platelets ≥ 100,000 cells/µl
* Women must have had last dose of chemotherapy at least 3 weeks prior to treatment with PVSRIPO
* Women must have at least 2 weeks minimum (ideal 3-4 weeks) of a wash-out period after any steroid administration (IV, PO, or intraocular)
* Serum creatinine ≤ 1.5 mg/dl, serum SGOT and bilirubin ≤ 1.5 times ULN (upper limit of normal)
* Women must provide written informed consent prior to enrollment on study, prior to conduct of screening procedures and enrollment on study
* Women of childbearing potential will have a negative serum pregnancy test at screening
* Women of childbearing potential must be willing to avoid pregnancy for the course of the study through 120 days after PVSRIPO injection
* Surgical resection of the tumor is planned and patient is willing to undergo surgical resection of the cancer

Exclusion Criteria:

* T1 N0 invasive breast cancer
* Breast cancer with skin necrosis
* Concurrent immune therapy, chemotherapy, or steroid therapy
* Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks prior to polio vaccine booster
* Has a known diagnosis of immunodeficiency
* Has a known additional malignancy that is progressing or requires active treatment
* Has known active central nervous system metastases and/or carcinomatous meningitis
* Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease or a syndrome that requires systemic steroids or immunosuppressive agents
* Has an active infection requiring systemic therapy
* Has known psychiatric or substance abuse disorders that would interfere with the requirements of the trial
* Is pregnant, breastfeeding, or expecting to conceive children within the projected duration of the trial, starting with the screening visit through 120 days after trial treatment
* Has received prior therapy with an anti-PD-1, anti-PDL-1, anti-PDL-2, anti-CD137, or anti-CTLA-4 (or any other antibody or drug specifically targeting T cell co-stimulation or checkpoint pathways)
* Has a known history of Human Immunodeficiency Virus (HIV)
* Has known active Hepatitis B or Hepatitis C
* Active liver disease with elevated transaminases > 2x ULN
* Has received a live vaccine within 30 days prior to PVSRIPO treatment

  * Inactivated vaccines are acceptable and are not an exclusion criterion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women
Enrollment: 5 (Actual)
Dates: Start 2019-06-30 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2022-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darell Bigner, MD, PhD, Study Director — Istari Oncology, Inc.
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants Treated: All participants received a single lerapolturev dose
Period: Overall Study
Arm/Group | All Participants Treated
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants Treated
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Tumor Infiltrating Immune Cells
Description: To describe the change in the amount of tumor infiltrating immune cells in tumor tissue pre- and post-injection of PVSRIPO
Time Frame: 10-20 days post-Injection of PVSRIPO
Population: participants tumor tissue available pre- and post-treatment with PVSRIPO
Measure: Mean (Standard Deviation); unit: fold-change of % CD45+ cells
Arm/Group | All Participants Treated
Number analyzed (Participants) | 3
fold-change of % CD45+ cells | 2.6 (1.3)

ADVERSE EVENTS:
Time Frame: From treatment until study discontinuation, an average of 5 months
Arm/Group | All Participants Treated
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 3/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants Treated (N=5)
COVID-19 infection (Infections and infestations) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Injection Site Reaction (General disorders) | 1 (1)
Aspartate Aminotransferase Increase (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-12): https://cdn.clinicaltrials.gov/large-docs/82/NCT03564782/Prot_SAP_000.pdf